CLINICAL TRIAL: NCT06460246
Title: Pulse Oximeter Accuracy During Stable Hypoxia Plateaus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acurable Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00077383
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulse Oximeter (Experimental): The subjects will have a 22-gauge catheter inserted in the radial artery to measure the oxygen saturation of arterial blood and also wear pulse oximeters.
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter — The subjects will have a 22-gauge catheter inserted in the radial artery to measure the oxygen saturation of arterial blood and also wear pulse oximeters.

SUMMARY:
This project aims to test the accuracy of pulse oximeters in the range of arterial HbO2 saturations from 100% down to 70%.

DETAILED DESCRIPTION:
This project aims to test the accuracy of pulse oximeters in the range of arterial HbO2 saturations from 100% down to 70%. This is done by comparing the pulse oximeter reading during brief, steady state hypoxia plateaus with a gold-standard measurement of blood oxyhaemoglobin saturation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged >= 18 and < 50.
* Subject in good general health with no evidence of any medical problems.
* Subject is fluent in both written and spoken English.
* Subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* Subject is obese (BMI > 35).
* Subject has a known history of heart disease, lung disease, kidney, or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* Subject has hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* Subject has any other serious systemic illness.
* Subject is a current smoker.
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators would interfere with the sensors working correctly.
* Subject has a history of fainting or vasovagal response.
* Subject has a history of sensitivity to local anesthesia.
* Subject has a diagnosis of Raynaud's disease.
* Subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* Subject is pregnant, lactating, or trying to get pregnant.
* Subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* Subject has any other condition, which in the opinion of the investigators would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Performance of the pulse oximeters against corresponding arterial blood oxygen saturation. | 1-4 hours
  Performance of the pulse oximeters against corresponding arterial blood oxygen saturation.

CONTACTS AND LOCATIONS:
Locations (1):
- Vital Signs Research Group, L.L.C., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No